CLINICAL TRIAL: NCT06691165
Title: Low Oxygen Therapy as a Cardiac Treatment for Improving 24-hour Blood Pressure Stability in Spinal Cord Injury
Brief Title: Improving 24-hour Blood Pressure Stability in Spinal Cord Injury With Low Oxygen Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glen Foster (Other)
Responsible Party: Sponsor-Investigator, Glen Foster, Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H24-02648; F23-01237 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-10-23; First posted 2024-11-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: Low oxygen therapy; Intermittent hypoxia; Blood pressure; Spinal cord injury; Cardiac function; Sympathetic nervous system
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Room air control; lot oxygen therapy; recovery/washout (Experimental): Participants with chronic cervical spinal cord injury will undergo a 4-day low oxygen therapy intervention.
  Measurements will first be taken at least three days before the beginning of the intervention to establish baseline characteristics, immediately before and after the first day of the intervention to assess the acute response to the intervention, and on the first and fourth days after the end of the intervention to assess persistent effects and washout.
  Interventions: Drug: Low oxygen therapy (LOT)

INTERVENTIONS:
Drug: Low oxygen therapy (LOT) — Participants will breathe variable concentrations of inspired oxygen, carbon dioxide, and nitrogen. The concentrations will be adjusted on a breath-by-breath basis to maintain end-tidal targets.
  Each daily session of the intervention will consist of forty 1-minute intervals. Each 1-minute interval will consist of 40 seconds of hypercapnic hypoxia, increasing the partial pressure of end-tidal carbon dioxide by +4 mmHg and decreasing the partial pressure of end-tidal oxygen to 45 mmHg, followed by 20 seconds in simulated room air to return to baseline carbon dioxide and oxygen levels.
  Other Names: Intermittent hypoxia

SUMMARY:
This study examines the effects of low oxygen therapy (LOT) on the stability of 24-hour blood pressure in persons with chronic cervical spinal cord injury.

This study will examine if brief episodes of breathing lower oxygen, termed low oxygen therapy (LOT), which has been shown to enhance autonomic nervous system activity, can improve blood pressure stability in individuals with spinal cord injury. The research team will assess 24-hour blood pressure, as well as cardiac, vascular, and autonomic function before and after a 4-day LOT treatment intervention. This study will advance current understanding of treatments to mitigate cardiovascular disease risk in people with spinal cord injuries.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) interrupts signals travelling down from the brain to the rest of the body below the level of the injury. The loss of nerve connections involved in cardiovascular control results in blood pressure instability. This can lead to sudden drops in blood pressure, such as when shifting upright or during transfers, or sudden increases during autonomic dysreflexia. These swings in blood pressure are linked to a nearly 4-fold increase in the risk of cardiovascular disease in people with SCI.

Repeated, brief exposure to breathing lower levels of oxygen, termed low oxygen therapy, has been shown to stimulate adaptation in the nervous system. This neuroplasticity increases the activity of cardiovascular control circuits, and has been shown to increase blood pressure in able-bodied individuals. Similar effects on respiratory and motor function in people with SCI, but the effects on the cardiovascular system have not been studied in this population.

This study will test the effects of a 4-day low oxygen therapy intervention on 24-hour blood pressure stability in people with chronic cervical SCI. By assessing mechanisms of cardiac, vascular, and autonomic function, this study aims to improve current understanding of the therapeutic potential of low oxygen therapy to mitigate cardiovascular disease risk in SCI.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 19-65
* Living with a chronic cervical (at or above T1) spinal cord injury of at least one year
* Are fluent in english

Exclusion Criteria:

* High-cervical injuries requiring ventilator assistance to breathe will be excluded on account of the necessity of the facemask for the delivery of hypoxia
* Unhealed fracture, contracture, or pressure sore that might interfere with participants' ability to complete the protocol
* Additional concurrent neurological conditions (e.g., multiple sclerosis, Parkinson disease, stroke or brain injury)
* Uncontrolled cardiovascular or pulmonary disease
* Severe neuropathic pain
* Severe recurrent autonomic dysreflexia
* History of seizure disorders
* Known pregnancy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour blood pressure | Change from baseline of 24-hour mean arterial blood pressure at 1-day post-intervention
  Mean arterial blood pressure (mmHg), averaged across 24 hours

SECONDARY OUTCOMES:
Change in 24-hour blood pressure stability | Change from baseline of the standard deviation of 24-hour mean arterial blood pressure at 1-day post-intervention
  Mean arterial blood pressure (mmHg), standard deviation across 24 hours
Change in left-ventricular contractility | Change from baseline of left ventricular contractility indices immediately after the first intervention session, and at 1-day and 4-days post-intervention
  Indices of load-independent pressure generation during systole: Estimated end-systolic elastance (mmHg/ml); end-systolic pressure-volume relationship slopes (mmHg/ml)
Change in baroreflex gain | Change from baseline of baroreflex gain indices immediately after first intervention session, and at 1-day and 4-days post-intervention
  Indices of baroreflex sensitivity: Relationship of systolic blood pressure against subsequent R-R interval duration during Valsalva Maneuver phases II and IV (ms/mmHg); spectral power of low-frequency resting blood pressure variability
Change in circulating catecholamines | Change from baseline of circulating catecholamines immediately after first intervention session, and at 1-day and 4-days post-intervention
  Venous plasma concentrations of norepinephrine and epinephrine (mmol/L)
Change in cerebral neurovascular coupling and autoregulation | Change from baseline of the responses of cerebral blood flow indices during a visual stimulus and head-up tilt immediately after first intervention session, and at 1-day and 4-days post-intervention
  Middle and posterior cerebral artery blood flow velocity (cm/s)
Change in renal filtration function | Change from baseline in renal biomarkers and blood flow at rest immediately after first intervention session, and at 1-day and 4-days post-intervention
  Humoral renal biomarkers (e.g., serum creatinine)
Change in flow-mediated dilation | Change from baseline in flow-mediated dilation immediately after first intervention session, and at 1-day and 4-days post-intervention
  Brachial artery flow-mediated dilation following 5-minute forearm blood flow occlusion (mm)
Change in tonic peripheral chemoreflex activity | Change from baseline in the magnitude of ventilatory depression in hyperoxia immediately after first intervention session, and at 1-day and 4-days post-intervention
  Magnitude of hyperoxic ventilatory depression (L/min)
Change in renal vascular function | Change in renal blood flow velocity from baseline during the first and final hypoxia cycles on the first session of the intervention
  Renal artery blood flow velocity (cm/s)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - UBC Okanagan, Kelowna, British Columbia
  - International Collaboration on Repair Discoveries (ICORD), Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vermeulen TD, Benbaruj J, Brown CV, Shafer BM, Floras JS, Foster GE. Peripheral chemoreflex contribution to ventilatory long-term facilitation induced by acute intermittent hypercapnic hypoxia in males and females. J Physiol. 2020 Oct;598(20):4713-4730. doi: 10.1113/JP280458. Epub 2020 Aug 19. PMID 32744340
- [Background] Claydon VE, Steeves JD, Krassioukov A. Orthostatic hypotension following spinal cord injury: understanding clinical pathophysiology. Spinal Cord. 2006 Jun;44(6):341-51. doi: 10.1038/sj.sc.3101855. Epub 2005 Nov 22. PMID 16304564
- [Background] Vose AK, Welch JF, Nair J, Dale EA, Fox EJ, Muir GD, Trumbower RD, Mitchell GS. Therapeutic acute intermittent hypoxia: A translational roadmap for spinal cord injury and neuromuscular disease. Exp Neurol. 2022 Jan;347:113891. doi: 10.1016/j.expneurol.2021.113891. Epub 2021 Oct 9. PMID 34637802
- [Background] Perim RR, Vinit S, Mitchell GS. Cervical spinal hemisection effects on spinal tissue oxygenation and long-term facilitation of phrenic, renal and splanchnic sympathetic nerve activity. Exp Neurol. 2023 Oct;368:114478. doi: 10.1016/j.expneurol.2023.114478. Epub 2023 Jul 13. PMID 37451584
- [Background] Welch JF, Vose AK, Cavka K, Brunetti G, DeMark LA, Snyder H, Wauneka CN, Tonuzi G, Nair J, Mitchell GS, Fox EJ. Cardiorespiratory Responses to Acute Intermittent Hypoxia in Humans With Chronic Spinal Cord Injury. J Neurotrauma. 2024 Sep;41(17-18):2114-2124. doi: 10.1089/neu.2023.0353. Epub 2024 Apr 18. PMID 38468543